CLINICAL TRIAL: NCT03576261
Title: Does Heart Failure Has Impact on Hemodynamic Stability During Anesthesia Induction
Brief Title: Heart Failure and Hemodynamic Stability During Anesthesia Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Tomi Myrberg, Principal investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016/361-31 III
Record Dates: First submitted 2018-06-04; First posted 2018-07-03 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Hemodynamic Instability; Anesthesia; Adverse Effect; Heart Failure; Diastolic Dysfunction; Venous; Return (Anomaly)
Keywords: hemodynamics; venous return; heart failure; anesthesia
MeSH Terms: conditions — Heart Failure; Congenital Abnormalities | interventions — Polygeline

STUDY DESIGN:
Intervention Model Description: A consecutive cohort. Signed informed consent is gathered. Non-blinded randomization is conducted to fluid therapy before anesthesia induction. Preoperative diagnostics by echocardiography is conducted to all participants.Two arms, with or without preoperative fluids, are studied regarding hemodynamic stability during anesthesia induction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative echo + fluids (Experimental): 20 individuals investigated by preoperative transthoracic echocardiography. Preoperative colloid fluid bolus (Gelofusine, Fresenius Kabi AB, Sweden) 6 ml/kg lean body weight, is infused intravenously immediately before anesthesia induction.
  Interventions: Other: Preoperative colloid fluid bolus (Gelofusine); Diagnostic Test: Preoperative transthoracic echocardiography
- Preoperative echo, control (Active Comparator): 20 individuals investigated by preoperative transthoracic echocardiography. No intravenous fluids are infused before anesthesia induction.
  Interventions: Diagnostic Test: Preoperative transthoracic echocardiography

INTERVENTIONS:
Other: Preoperative colloid fluid bolus (Gelofusine) — Preoperative colloid fluid bolus
  Arms: Preoperative echo + fluids
Diagnostic Test: Preoperative transthoracic echocardiography — Screening of biventricular systolic and diastolic function of the heart and level of venous return by transthoracic echocardiography approximately one hour before preoperative fluid therapy and anesthesia induction.

SUMMARY:
The study aim is to investigate whether preoperative heart failure has impact on hemodynamic stability during anesthesia induction by target controlled infusion of anesthesia (TCI) in non-cardiac, non-morbidly obese surgery.

DETAILED DESCRIPTION:
40 individuals are enrolled to the study after signed informed consent at the day of surgery. The study participants are randomized (non-blinded) to preoperative fluid therapy (preoperative colloid fluid bolus at 6 ml/kg LBW, Gelofusine™, Fresenius Kabi AB, Sweden) or control (no preoperative fluids) before standardized TCI- induction of anesthesia. No other intravenous fluids before anesthesia induction.

Preoperative screening of biventricular systolic and diastolic function of the heart and level of venous return is implemented by transthoracic echocardiography approximately one hour before preoperative fluid therapy and anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* body mass index ≤ 35 kg/m2
* electively scheduled for breast cancer surgery, endocrinologic surgery (thyroid, parathyroid) and general abdominal surgery

Exclusion Criteria:

* instable angina pectoris
* severe bronchial asthma
* severe COPD
* dementia
* severe heart valve disease
* severe renal failure
* body mass index > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of blood pressure drops | 20 minutes post anesthesia induction
  Blood pressure drop below mean arterial pressure at 65 mmHg during anesthesia induction. Non-invasive blood pressures (systolic, mean and diastolic) are measured 5 minutes before anesthesia induction and thereafter every 5 minutes post-induction .
Incidence of severe blood pressure drops | 20 minutes post anesthesia induction
  Blood pressure drop below mean arterial pressure at 55 mmHg during anesthesia induction. Non-invasive blood pressures (systolic, mean and diastolic) are measured 5 minutes before anesthesia induction and thereafter every 5 minutes post-induction.

SECONDARY OUTCOMES:
Venous return and hemodynamic stability | 20 minutes post anesthesia induction
  Level of venous return impact on blood pressure drops during anesthesia below mean arterial pressure at 65 mmHg
Systolic heart failure and hemodynamic stability | 20 minutes post anesthesia induction
  Systolic heart failure impact on blood pressure drops during anesthesia below mean arterial pressure at 65 mmHg
Diastolic dysfunction and hemodynamic stability | 20 minutes post anesthesia induction
  Diastolic dysfunction impact on blood pressure drops during anesthesia below mean arterial pressure at 65 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Tomi Myrberg, MD PhD, Principal Investigator — Umea Universitet
Locations (1):
- Sunderby teaching hospital, Luleå, Sweden

IPD SHARING:
Plan to Share IPD: No